CLINICAL TRIAL: NCT00778349
Title: A Randomized, Three-Treatment, Three-Period, Six-Sequence, Single-Dose, Crossover Pharmacokinetic Study on Metformin Hydrochloride Solution 100 mg/mL of Ranbaxy Laboratories Comparing the Pharmacokinetic Profile of Metformin Under Fasting Condition, After a Low Fat Meal and After a High Fat Meal in Healthy, Adult, Human Male Subjects.
Brief Title: A Comparitive Bioavailability Study of Metformin Hydrochloride Liquid 500mg/ 5 mL Under Fasting Conditions and After Low and High Fat Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 04/METFO-500/02
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioavailability Metformin solution 100 mg/mL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Metformin solution 100 mg/mL under fasting condition
  Interventions: Drug: Metformin solution 100 mg/mL
- 2 (Experimental): Metformin solution 100 mg/mL, after low fat meal
  Interventions: Drug: Metformin solution 100 mg/mL
- 3 (Experimental): Metformin solution 100 mg/mL, after high fat meal
  Interventions: Drug: Metformin solution 100 mg/mL

INTERVENTIONS:
Drug: Metformin solution 100 mg/mL

SUMMARY:
To assess the food effect on pharmacokinetic profile of metformin liquid 100 mg/mL of Ranbaxy Laboratories in healthy, adult, human subjecis following a dose administration of 10 mL (1000 mg) under fasting conditions, after a Iow fat meal and after a high fat meal

DETAILED DESCRIPTION:
This study was an open label, randomized, three-treatment, three-period, six-sequence, single-dose, crossover pharmacokinetic study planned on 36 healthy, adult, human subjects under fasting conditions. However 34 subjects were enrolled and 33 subjects completed all the periods of the study. All periods were separated by a washout of seven days As per protocol (Appendix 1), enough healthy, adult, human subjects were to be enrolled in the study to allow the dosing of 36 subjects in the first period. 34 subjects were enrolled and 33 subjects completed all the periods of study

ELIGIBILITY:
Inclusion Criteria:

1. Be in the age range of 18.45 years.
2. Be neither overweight nor underweight for his/her height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Have voluntarily given written informed consent to participate in this study.
4. Be of normal health as determined by medical history and physical
5. Examination of the subjects performed .within 28 days prior to the commencement of the study.
6. If female and:

Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or~ Is postmenopausal for at least 1 year; or Is surgically sterile bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

1. History of allergy to metformin and other related antidiabetic biguanide preparations.
2. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
3. Presence of disease markers of HIV 1 and 2, Hepatitis B and C viruses and syphilis infection.
4. Female volunteers demonstrating a positive pregnancy screen.
5. Female volunteers who are currently breastfeeding.
6. Presence of values' which are clinically significantly different from normal reference ranges for hemoglobin, total white blood cells count, differential WBC count and platelet count
7. Positive for urinary screen testing of drugs of abuse (opiates and cannabinoids
8. Presence of values which are significantly different from normal.reference ranges (as defined in Appendix 5) for se- rum creatinine, blood urea nitrogen serum aspartate aminotransferase (AST), serum alanine aminotranferase (ALT), serum alkaline phosphatase, serum billrubin, plasma glucose and serum cholesterol
9. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose, (positive) and protein (positive).
10. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes or glaucoma.
11. History of any psychiatric illness. which may impair the ability to provide written informed consent.
12. Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
13. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 'unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
14. Use of any enzyme modifying drugs within 30 days prior to Day I of this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2002-04; Primary Completion 2002-05 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Bioavailability

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html